CLINICAL TRIAL: NCT04026945
Title: A Dose-Escalating Phase I Study of a Single Injection of Lidocaine Paste (ST-CP) for Spermatic Cord Block in Men With Chronic Scrotal Content Pain
Brief Title: Sustained Release Lidocaine for Treatment of Scrotal Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ryan Flannigan, MD, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H19-00438
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pain
Keywords: chronic scrotal pain; chronic testicular pain; spermatic cord; orchialgia; chronic scrotal content pain
MeSH Terms: conditions — Chronic Pain | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Treatment (ST-CP) Group (Other): This study uses a dose-escalating approach in the active treatment arm. There is no comparator product. All qualifying patients receive the active treatment ST-CP as an injection in the region around the spermatic cord. The following dosing cohorts will be used:
  I: 1 x 2 mL of 140 mg/mL ST-CP (= 280 mg lidocaine) II: 1 x 3 mL of 140 mg/mL ST-CP (= 420 mg lidocaine) III: 1 x 4 mL of 140 mg/mL ST-CP (= 560 mg lidocaine)
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Sustained-release lidocaine injection
  Other Names: ST-CP Lidocaine; ST-CP; Sustained-release lidocaine

SUMMARY:
In this study, the investigators are testing a new formulation of lidocaine for its suitability in managing chronic scrotal pain (CSCP). The new formulation ST-CP is a lidocaine sustained-release formulation and is expected to provide pain relief over 4 weeks. Currently, the drug lidocaine is not available as an injectable slow-release formulation and chronic scrotal pain patients are often left untreated.

DETAILED DESCRIPTION:
The purpose of this study is to find out if a new polymeric, water-free formulation of lidocaine is safe and can provide effective, long-lasting pain relief in chronic scrotal pain (CSCP) patients. This new formulation ST-CP is injected into the spermatic cord of patients in a very comparable way that the currently available lidocaine solution (Lidocaine HCl 1% USP) is administered. The only difference is that the polymer solution stays in the area of injection longer by forming a soft implant.

The investigators therefore hypothesize that the polymer formulation of lidocaine will release the drug over an extended period of time and will not dissolve away like the currently used lidocaine solution (Lidocaine HCl 1%, USP). This will lead to long-lasting pain relief for CSCP patients.

The investigators' primary objective is to determine if the single injection of our polymeric lidocaine formulation is well tolerated by patients with CSCP. Secondary objectives are to determine the duration and extent of pain relief, the impact of ST-CP on pain-related quality of life and the systemic exposure to lidocaine.

The clinical study is conducted at the Vancouver Prostate Centre. Potential participants will undergo a screening period to determine basal pain levels over 7 days and test their ability to respond to a spermatic cord block with a standard lidocaine injection (Lidocaine HCl 1%, USP). Up to 15 men will receive our ST-CP study formulation and will be monitored over the the following 4 weeks. Follow-up procedures will include blood draws, daily pain evaluations and standard questionnaires on scrotal pain and erectile function. Up to 3 dose levels are planned but dose escalation will only occur once the previous cohort (3 patients) has completed the follow up and safety assessment.

Summary descriptive statistics (including mean and standard deviation, median, range, proportion) will be provided for important parameters and outcome measures. These include subject demographics, subject disposition, subject compliance, pharmakokinetic laboratory test outcomes, overall adverse events, adverse events related to lidocaine and adverse events related to study procedure. Pain scores and questionnaires will be summarized by score and pre- and post- treatment levels will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Adult ( ≥ 19 years) male
* Unilateral scrotal pain lasting >3 months
* Average daily maximum scrotal pain score over 7 days ≥ 5 on the 0-10 NRS (see study protocol attached in 9.1.)
* Positive response to test spermatic cord block with 1% Lidocaine (Lidocaine HCl 1%, USP), defined as a temporary decrease of at least two points on the NRS (see study protocol attached in 9.1.) within an hour of injection

Exclusion Criteria:

* Negative response to test spermatic cord block, defined as absence of a temporary decrease of at least two points on the NRS (see study protocol attached in 9.1.) within an hour of injection
* Other pain generator site with NRS ≥ 5
* History of allergic reaction to lidocaine or any other component of ST-CP Lidocaine
* Known hypersensitivity to anesthetics of the amide-type.
* Complete heart block.
* Use of anticoagulants (Aspirin permitted)
* Active infection involving the urinary tract or scrotum
* Inability to give consent
* Inability to follow up according to the protocol
* Negative response to previous spermatic cord block.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 28 days
  Determination of safety and tolerability of the study treatment ST-CP through the assessment of adverse events

SECONDARY OUTCOMES:
NRS Pain Score | 28 days
  Determination of daily maximum pain score over 14 and 28 days
Validated Chronic Epididymitis Symptom Index (CESI) | 28 days
  Determination of the pain associated quality of life
Validated International Index of Erectile Function (IIEF-5) | 28 days
  Determination of erectile function associated quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Flannigan, MD, Principal Investigator — University of British Columbia; Ryan Paterson, MD, Principal Investigator — University of British Columbia
Locations (1):
- Department of Urologic Sciences, Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia, Canada